CLINICAL TRIAL: NCT03413735
Title: Dietary Green Tea Confection For Resolving Gut Permeability-Induced Metabolic Endotoxemia In Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Richard Bruno, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017H0246
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Endotoxemia; Inflammation
MeSH Terms: conditions — Obesity; Endotoxemia; Inflammation | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Confection (Placebo Comparator): Confection without green tea extract consumed daily for 4 weeks
  Interventions: Other: Placebo
- Green Tea Extract-Confection (Experimental): Confection with green tea extract consumed daily for 4 weeks
  Interventions: Other: Green Tea Extract

INTERVENTIONS:
Other: Green Tea Extract — Confections containing green tea extract that will be ingested daily for 4 weeks
  Arms: Green Tea Extract-Confection
Other: Placebo — Confections containing no green tea extract that will be ingested daily for 4 weeks
  Arms: Placebo Confection

SUMMARY:
This study is focused on assessing gastrointestinal-level improvements by which green tea limits metabolic endotoxemia. It is completed in two phases. Phase I consists of a pharmacokinetic study to examine the bioavailability of green tea catechins among lean and obese persons who consumed a single dose of a green tea extract (GTE)-containing confection. These persons will then complete phase 2, which consists of a parallel design randomized controlled in which lean and obese persons will consume placebo or GTE confections.

It is expected that catechin-rich green tea will improve gut barrier function to prevent endotoxin translocation and associated low-grade inflammation. Outcomes will therefore support dietary recommendations for green tea to alleviate obesity-related inflammatory responses. Specifically, the study is expected to demonstrate that a green tea confection snack food can attenuate metabolic endotoxemia in association with restoring gastrointestinal health.

DETAILED DESCRIPTION:
Obesity is a major public health concern in the United States, with over two-thirds of the adult population classified as overweight or obese. Obesity is characterized by low-grade chronic inflammation that, in part, is mediated by metabolic endotoxemia. Metabolic endotoxemia describes increased circulating levels of gut-derived endotoxin (a bacterial product derived from Gram-negative bacteria in the intestines) that results from gut barrier dysfunction, a phenomenon that is common in obesity. Studies in rodents models have shown that dietary supplementation with green tea extract (GTE) reduces metabolic endotoxemia in association with improved gut health. This clinical trial will therefore investigate the extent to which a green tea confection snack food can alleviate metabolic endotoxemia and restore gut health in obese humans. It is hypothesized that 4-week daily ingestion of a green tea extract (GTE)-rich confection will limit metabolic endotoxemia by decreasing gut barrier permeability. This study will address the following objectives: 1) define alterations in catechin pharmacokinetics in obese compared with healthy adults, 2) demonstrate improvements in gut barrier function by GTE, and 3) demonstrate GTE-mediated amelioration of microbial dysbiosis.

To test the hypothesis, all participants will initially complete a 12-h pharmacokinetics study to define the influence of obesity on catechin bioavailability and metabolism. They will then be randomized to complete a double-blind, randomized, placebo-controlled trial where they will receive a GTE-rich or placebo confection for 4 weeks. Prior to and upon completing the intervention, participants will undergo a gut permeability test, fecal samples will be collected for microbiota composition analysis, and blood samples will be collected to assess endotoxin and inflammatory biomarkers. Upon successfully completing this study, it is anticipated that chronic consumption of a green tea confection will be demonstrated to be an effective dietary strategy to reduce metabolic endotoxemia and improve gut health.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese (BMI = 28-40 kg/m2)
* Fasting glucose < 126 mg/dL
* Normotensive (blood pressure < 140/90 mmHg)
* Non-dietary supplement user
* Non-smoker

Exclusion Criteria:

* Regular tea drinkers (> 2 cups/week)
* Vegetarians
* Use of medications to manage diabetes, hypertension, or hyperlipidemia
* Use of any medications known to be contraindicated for use with green tea ingestion
* User of dietary supplements, prebiotics, or probiotics
* Recent use of antibiotics or anti-inflammatory agents
* Women who are pregnant or lactating or have initiated or changed birth control in the past 3-months
* Individuals with gastrointestinal disorders or surgeries
* Individuals with hemochromatosis
* Alcohol intake > 3 drinks per day
* Any history of cancer

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bruno, PhD, RD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data will be published as aggregate only. Data sharing may be possible pending institutional agreements.

REFERENCES:
- [Background] Li J, Sapper TN, Mah E, Moller MV, Kim JB, Chitchumroonchokchai C, McDonald JD, Bruno RS. Green tea extract treatment reduces NFkappaB activation in mice with diet-induced nonalcoholic steatohepatitis by lowering TNFR1 and TLR4 expression and ligand availability. J Nutr Biochem. 2017 Mar;41:34-41. doi: 10.1016/j.jnutbio.2016.12.007. Epub 2016 Dec 21. PMID 28038359
- [Background] Li J, Sasaki GY, Dey P, Chitchumroonchokchai C, Labyk AN, McDonald JD, Kim JB, Bruno RS. Green tea extract protects against hepatic NFkappaB activation along the gut-liver axis in diet-induced obese mice with nonalcoholic steatohepatitis by reducing endotoxin and TLR4/MyD88 signaling. J Nutr Biochem. 2018 Mar;53:58-65. doi: 10.1016/j.jnutbio.2017.10.016. Epub 2017 Nov 3. PMID 29190550

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Phase 1, participants were stratified by phenotype (lean vs. obese) and received a single dose of a green tea extract (GTE)-enriched confection. This phase was conducted to evaluate catechin bioavailability. All participants consumed the same GTE confection. After a washout period, participants were randomized in Phase 2 to receive either a GTE or placebo confection daily for 4 weeks in a double-blind trial.
Groups:
- Lean - Placebo; Obese - Placebo: Confection without green tea extract consumed daily for 4 weeks
  Placebo: Confections containing no green tea extract that will be ingested daily for 4 weeks
- Lean - GTE; Obese - GTE: Confection with green tea extract consumed daily for 4 weeks
  Green Tea Extract: Confections containing green tea extract that will be ingested daily for 4 weeks
Period: Pharmacokinetic Study
Arm/Group | Lean - Placebo | Lean - GTE | Obese - Placebo | Obese - GTE
Started (All participants in this arm received a single dose of GTE in Phase 1. This arm label reflects phenotype and randomized group assignment for Phase 2 only.) | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Randomized Controlled Trial
Arm/Group | Lean - Placebo | Lean - GTE | Obese - Placebo | Obese - GTE
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 9 | 10
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Confection | Green Tea Extract-Confection | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28. (6.48) | 28.35 (9.04) | 28.175 (7.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 8 | 12 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Endotoxin
Description: Serum endotoxin concentration
Time Frame: Week 0 - Fasting
Measure: Mean (Standard Deviation); unit: EU/mL
Groups:
- Lean - GTE; Obese - GTE: Participants consumed green tea extract containing confection (50 g 114 confection containing 0.5 g GTE) without any additional foods, except water (500 mL).
- Lean - Placebo; Obese - Placebo: Participants consumed gelatin extract with no green tea extract.
Arm/Group | Lean - GTE | Obese - GTE | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
EU/mL | 14.44 (4.46) | 12.97 (6.44) | 12.25 (6.05) | 17.65 (12.58)

2. Primary Outcome: Endotoxin
Description: Serum endotoxin concentration
Time Frame: Week 2 - Fasting
Measure: Mean (Standard Deviation); unit: EU/mL
Arm/Group | Lean - GTE | Obese - GTE | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
EU/mL | 13.59 (7.38) | 12.38 (7.53) | 13.00 (5.44) | 15.62 (5.32)

3. Primary Outcome: Endotoxin
Description: Serum endotoxin concentration
Time Frame: Week 4 - Fasting
Measure: Mean (Standard Deviation); unit: EU/mL
Groups:
- Lean; Obese: Participants consumed green tea extract containing confection (50 g 114 confection containing 0.5 g GTE) without any additional foods, except water (500 mL).
Arm/Group | Lean | Obese | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
EU/mL | 12.33 (4.55) | 16.46 (4.91) | 11.33 (5.56) | 15.45 (6.94)

4. Secondary Outcome: Gut Permeability - Lactulose to Mannitol Ratio
Description: Urinary Lactulose/Mannitol Ratio (mg/mg)
Time Frame: Week 0 - 0-5 hours
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Lean - Placebo; Obese - Placebo: Participants consumed a gelatin confection that did not contain green tea extract.
Arm/Group | Lean - GTE | Obese - GTE | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9
Ratio | 0.12 (0.06) | 0.09 (0.03) | 0.10 (0.05) | 0.10 (0.03)

5. Secondary Outcome: Gut Permeability - Lactulose to Mannitol Ratio
Description: Urinary Lactulose/Mannitol Ratio (mg/mg)
Time Frame: Week 0 - 6-24 hours
Measure: Mean (Standard Deviation); unit: Urinary Lactulose/Mannitol Ratio (mg/mg)
Groups:
- Lean - Placebo; Obese - Placebo: Participants consumed a gelatin confection with no green tea extract.
Arm/Group | Lean - GTE | Obese - GTE | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9
Urinary Lactulose/Mannitol Ratio (mg/mg) | 0.16 (0.10) | 0.11 (0.10) | 0.19 (0.12) | 0.19 (0.14)

6. Secondary Outcome: Gut Permeability - Lactulose to Mannitol Ratio
Description: Urinary Lactulose/Mannitol Ratio (mg/mg)
Time Frame: Week 4 - 0-5 hours
Measure: Mean (Standard Deviation); unit: Urinary Lactulose/Mannitol Ratio (mg/mg)
Arm/Group | Lean - GTE | Obese - GTE | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9
Urinary Lactulose/Mannitol Ratio (mg/mg) | 0.12 (0.13) | 0.14 (0.10) | 0.10 (0.06) | 0.12 (0.08)

7. Secondary Outcome: Gut Permeability - Lactulose to Mannitol Ratio
Description: Urinary Lactulose/Mannitol Ratio (mg/mg)
Time Frame: Week 4 - 6-24 hours
Measure: Mean (Standard Deviation); unit: Urinary Lactulose/Mannitol Ratio (mg/mg)
Arm/Group | Lean - GTE | Obese - GTE | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9
Urinary Lactulose/Mannitol Ratio (mg/mg) | 0.14 (0.11) | 0.18 (0.18) | 0.19 (0.12) | 0.21 (0.12)

8. Secondary Outcome: Gut Permeability - Sucralose to Erythritol Ratio
Description: Urinary Sucralose/Erythritol Ratio (mg/mg)
Time Frame: Week 0 - 6-24 hours
Measure: Mean (Standard Deviation); unit: Urinary Sucralose/Erythritol (mg/mg)
Arm/Group | Lean - GTE | Obese - GTE | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9
Urinary Sucralose/Erythritol (mg/mg) | 0.02 (0.01) | 0.02 (0.01) | 0.02 (0.01) | 0.02 (0.01)

9. Secondary Outcome: Gut Permeability - Sucralose to Erythritol Ratio
Description: Urinary Sucralose/Erythritol Ratio (mg/mg)
Time Frame: Week 0 - 0-24 hours
Measure: Mean (Standard Deviation); unit: Urinary Sucralose/Erythritol (mg/m
Arm/Group | Lean - GTE | Obese - GTE | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9
Urinary Sucralose/Erythritol (mg/m | 0.02 (0.01) | 0.02 (0.01) | 0.02 (0.004) | 0.02 (0.004)

10. Secondary Outcome: Urinary Sucralose/Erythritol Ratio (mg/mg)
Description: Ratio of excretion of urinary sugars (Sucralose to Erythritol)
Time Frame: Week 4 - 6-24 hours
Measure: Mean (Standard Deviation); unit: Urinary Sucralose/Erythritol (mg/m
Arm/Group | Lean - GTE | Obese - GTE | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9
Urinary Sucralose/Erythritol (mg/m | 0.01 (0.01) | 0.01 (0.01) | 0.02 (0.01) | 0.02 (0.02)

11. Secondary Outcome: Gut Permeability - Sucralose to Erythritol Ratio
Description: Urinary Sucralose/Erythritol Ratio (mg/mg)
Time Frame: Week 4 - 0-24 hours
Measure: Mean (Standard Deviation); unit: Urinary Sucralose/Erythritol (mg/m
Arm/Group | Lean - GTE | Obese - GTE | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9
Urinary Sucralose/Erythritol (mg/m | 0.01 (0.02) | 0.02 (0.01) | 0.02 (0.01) | 0.02 (0.01)

12. Secondary Outcome: Firmicutes to Bacteroidetes Ratio - Microbiota
Description: Ratio of fecal relative Firmicutes (% abundance)/Bacteroidetes (% abundance)
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: % of abundance
Arm/Group | Lean - GTE | Obese - GTE | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9
% of abundance | 4.34 (3.17) | 3.52 (2.32) | 21.51 (31.65) | 9.36 (7.48)

13. Secondary Outcome: Firmicutes to Bacteroidetes Ratio - Microbiota
Description: Ratio of fecal relative Firmicutes (% abundance)/Bacteroidetes (% abundance)
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lean - GTE | Obese - GTE | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9
ratio | 4.90 (3.74) | 8.95 (15.13) | 4.69 (4.17) | 9.32 (3.95)

14. Secondary Outcome: Bioavailability - Epigallocatechin Gallate
Description: Area under the curve (AUC) of plasma epigallocatechin calculated from blood collected at 0, 0.25, 0.5, 1, 2, 3, 5, 8, 10, 12 hours post-ingestion of green tea confection. Epigallocatechin gallate is measured in umol/L over time (hours) resulting in the AUC.
Time Frame: Prior to intervention enrollment...0-12 hours post-ingestion of a green tea confection
Population: A pharmacokinetics study was completed regarding catechin bioavailability in all participants prior to the intervention randomization of treatment (GTE/Placebo). During this phase, all lean and obese participants of both groups consumed green tea extract containing confection. Bioavailability measures were then performed.
Measure: Mean (Standard Error); unit: umol/L x h
Arm/Group | Lean | Obese
Number analyzed (Participants) | 19 | 17
umol/L x h | 3.46 (0.3) | 2.62 (0.3)

15. Secondary Outcome: Bioavailability - Epigallocatechin
Description: Area under the curve (AUC) of plasma epigallocatechins calculated from blood collected at 0, 0.25, 0.5, 1, 2, 3, 5, 8, 10, 12 hours post-ingestion of green tea confection. Epigallocatechin is measured in umol/L over time (hours) resulting in the AUC.
Time Frame: Prior to intervention enrollment...0-12 hours post-ingestion of a green tea confection
Population: as for outcome 14
Measure: Mean (Standard Error); unit: umol/L x h
Arm/Group | Lean | Obese
Number analyzed (Participants) | 19 | 17
umol/L x h | 1.18 (0.1) | 0.88 (0.1)

16. Secondary Outcome: Bioavailability - Epicatechin Gallate
Description: Area under the curve (AUC) of plasma epicatechins calculated from blood collected at 0, 0.25, 0.5, 1, 2, 3, 5, 8, 10, 12 hours post-ingestion of green tea confection. Epicatechins is measured in umol/L over time (hours) resulting in the AUC.
Time Frame: Prior to the intervention enrollment...0-12 hours post-ingestion of a green tea confection
Population: as for outcome 14
Measure: Mean (Standard Error); unit: umol/L x h
Arm/Group | Lean | Obese
Number analyzed (Participants) | 19 | 17
umol/L x h | 1.06 (0.1) | 0.78 (0.1)

17. Secondary Outcome: Bioavailability - Epicatechin
Description: Area under the curve (AUC) of plasma epicatechins calculated from blood collected at 0, 0.25, 0.5, 1, 2, 3, 5, 8, 10, 12 hours post-ingestion of green tea confection. Epicatechin is measured in umol/L over time (hours) resulting in the AUC.
Time Frame: Prior to intervention enrollment...0-12 hours post-ingestion of a green tea confection
Population: as for outcome 14
Measure: Mean (Standard Error); unit: umol/L x h
Arm/Group | Lean | Obese
Number analyzed (Participants) | 19 | 17
umol/L x h | 0.78 (0.1) | 0.57 (0.04)

18. Secondary Outcome: Cmax of Epigallocatechin Gallate
Description: Maximum plasma concentration of catechins calculated from blood collected at 0, 0.25, 0.5, 1, 2, 3, 5, 8, 10, 12 hours post-ingestion of green tea confection
Time Frame: Prior to intervention enrollment...0-12 hours post-ingestion of green tea confection
Population: as for outcome 14
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Lean | Obese
Number analyzed (Participants) | 19 | 17
umol/L | 0.5 (0.04) | 0.38 (0.03)

19. Secondary Outcome: Cmax of Epigallocatechin
Description: as for outcome 18
Time Frame: Prior to intervention enrollment...0-12 hours post-ingestion of green tea confection
Population: as for outcome 14
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Lean | Obese
Number analyzed (Participants) | 19 | 17
umol/L | 0.22 (0.01) | 0.18 (0.01)

20. Secondary Outcome: Cmax of Epicatechin Gallate
Description: as for outcome 18
Time Frame: Prior to intervention enrollment...0-12 hours post-ingestion of green tea confection
Population: as for outcome 14
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Lean | Obese
Number analyzed (Participants) | 19 | 17
umol/L | 0.14 (0.01) | 0.09 (0.01)

21. Secondary Outcome: Cmax of Epicatechin
Description: as for outcome 18
Time Frame: Prior to intervention enrollment...0-12 hours post-ingestion of green tea confection
Population: as for outcome 14
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Lean | Obese
Number analyzed (Participants) | 19 | 17
umol/L | 0.16 (0.1) | 0.13 (0.1)

22. Secondary Outcome: Tmax of Epigallocatechin Gallate
Description: Time to maximal plasma concentration of catechins calculated from blood collected at 0, 0.25, 0.5, 1, 2, 3, 5, 8, 10, 12 hours post-ingestion of green tea confection
Time Frame: Prior to intervention enrollment...0-12 hours post-ingestion of green tea confection
Population: as for outcome 14
Measure: Mean (Standard Error); unit: h
Arm/Group | Lean | Obese
Number analyzed (Participants) | 19 | 17
h | 3.32 (0.25) | 2.65 (0.26)

23. Secondary Outcome: Tmax of Epigallocatechin
Description: as for outcome 22
Time Frame: Prior to intervention enrollment...0-12 hours post-ingestion of green tea confection
Population: as for outcome 14
Measure: Mean (Standard Error); unit: h
Arm/Group | Lean | Obese
Number analyzed (Participants) | 19 | 17
h | 1.92 (0.25) | 1.41 (0.15)

24. Secondary Outcome: Tmax of Epicatechin Gallate
Description: as for outcome 22
Time Frame: Prior to intervention enrollment...0-12 hours post-ingestion of green tea confection
Population: as for outcome 14
Measure: Mean (Standard Error); unit: h
Arm/Group | Lean | Obese
Number analyzed (Participants) | 19 | 17
h | 4.05 (0.24) | 3.94 (0.39)

25. Secondary Outcome: Tmax of Epicatechin
Description: as for outcome 22
Time Frame: Prior to intervention enrollment...0-12 hours post-ingestion of green tea confection
Population: as for outcome 14
Measure: Mean (Standard Error); unit: h
Arm/Group | Lean | Obese
Number analyzed (Participants) | 19 | 17
h | 1.66 (0.24) | 1.53 (0.19)

26. Secondary Outcome: Calprotectin
Description: Fecal calprotectin concentration
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: ug/g
Arm/Group | Lean - GTE | Obese - GTE | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
ug/g | 64.99 (79.07) | 27.54 (20.58) | 32.01 (25.52) | 62.62 (90.84)

27. Secondary Outcome: Calprotectin
Description: Fecal calprotectin concentration
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: ug/g
Arm/Group | Lean - GTE | Obese - GTE | Lean - Placebo | Obese - Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
ug/g | 249.62 (590.21) | 25.74 (13.94) | 36.20 (24.15) | 73.04 (103.90)

ADVERSE EVENTS:
Time Frame: 1 month
Description: Consumption of the formulated green tea extract did not put any of the participants at risk for serious adverse events, not did it put any participants at risk for all-cause omrtality.
Groups:
- Lean - Placebo: Lean Participants consumed a placebo confection for 1-month
- Obese - Placebo: Obese Participants consumed a placebo confection for 1-month
- Lean - GTE: Lean Participants consumed green tea extract containing confection (50 g 114 confection containing 0.5 g GTE) for 1-month
- Obese - GTE: Obese Participants consumed green tea extract containing confection (50 g 114 confection containing 0.5 g GTE) for 1-month
Arm/Group | Lean - Placebo | Obese - Placebo | Lean - GTE | Obese - GTE
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT03413735/Prot_SAP_000.pdf